CLINICAL TRIAL: NCT06483165
Title: F.A.S.T.-BE FAST Consumer Stroke Warning Signs Study
Brief Title: F.A.S.T.-BE FAST Stroke Warning Signs Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00077822
Record Dates: First submitted 2024-04-25; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A randomized parallel 2-group design will be used to allow a rigorous assessment of the comparative efficacy of the two acronyms (BE FAST and F.A.S.T.) among English-speaking adults of diverse race and ethnicity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BE FAST Group (Experimental): The experimental BE FAST acronym education messaging, including 5 stroke warning signs and a call-to-action to call 911, will be shown to the participants using a brief video.
  Interventions: Other: BE FAST Educational video
- F.A.S.T. Group (Active Comparator): The comparator F.A.S.T. acronym education messaging, including 3 stroke warning signs and a call-to-action to call 911, will be shown to the participants using a brief video.
  Interventions: Other: F.A.S.T. Educational Video

INTERVENTIONS:
Other: BE FAST Educational video — A 1-minute educational video format using BE FAST. Each acronym will be visually displayed in the video and audio voice over of each letter and corresponding phrase will be audible in English. The look, feel, and messaging in each video will be the same except for the acronyms.
  Arms: BE FAST Group
Other: F.A.S.T. Educational Video — A 1-minute educational video format using F.A.S.T. Each acronym will be visually displayed in the video and audio voice over of each letter and corresponding phrase will be audible in English. The look, feel, and messaging in each video will be the same except for the acronyms.
  Arms: F.A.S.T. Group

SUMMARY:
The goal of this randomized controlled trial is to learn whether the BE FAST (Balance, Eyes, Face, Arm, Speech, and Time) acronym works at least as well or better than the F.A.S.T. (Face drooping, Arm weakness, Speech difficulty, Time to call 911) acronym in helping participants learn and remember the warning signs of a stroke. The main questions it aims to answer are:

* Does the BE FAST acronym increase understanding among participants that calling 911 is the right first step they should take if a stroke is suspected?
* Does the BE FAST acronym perform as well as or better than the F.A.S.T. acronym in helping participants remember stroke warning signs on a letter-aided open-ended basis? Researchers will compare the BE FAST acronym to the F.A.S.T. acronym to see if the BE FAST acronym works at least as well as the F.A.S.T. acronym in teaching participants about the warning signs of a stroke and the importance of calling 911 if they suspect a stroke.

Participants will:

* Take a survey about their knowledge of stroke and its symptoms
* Watch a short video about one of the acronyms and then answer more questions about what they learned
* Take another survey after 30 days about the acronym they learned about

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent;
* Have access to a computer, tablet or mobile device with internet services;
* Proficient in reading and writing the English language; and
* Reside outside a medical facility.

Exclusion Criteria:

* Not able to provide written informed consent;
* Do not have access to a computer, tablet or mobile device with internet;
* Not proficient in reading and writing in English language; or
* Reside in a medical facility.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Intent to Call 911 30-Days Post Education | 30 days
  The identification of calling 9-1-1 as the accurate immediate action to stroke being suspected at 30-days post-educational intervention. Outcome is not being reported on a scale. We are using dichotomous coding of correct or incorrect response, with the response of "Call 9-1-1" being the correct response from the pick list.

SECONDARY OUTCOMES:
Warning Signs Net Positive Accuracy Score 30-Days Post Education | 30 days
  Net positive accuracy score on the common letters (symptoms) in both acronyms on a letter-aided open-ended basis at 30-days post-educational intervention. Outcome is not being reported on a scale. We are using dichotomous coding for the letters in each acronym, where 0 = completely incorrect and 1 = fully correct (i.e. higher scores mean a better outcome).

OTHER OUTCOMES:
Intent to Call 911 Immediately Post-Education | Immediately after intervention
  The identification of calling 9-1-1 as the accurate immediate action to stroke being suspected immediately following the educational intervention. Outcome is not being reported on a scale. We are using dichotomous coding of correct or incorrect response, with the response of "Call 9-1-1" being the correct response from the pick list.
Change in Warning Signs Net Positive Accuracy Score Immediately Post-Education | Immediately after intervention
  Net positive accuracy score on the common letters (symptoms) in both acronyms on a letter-aided open-ended basis immediately following the educational intervention. Outcome is not being reported on a scale. We are using dichotomous coding for the letters in each acronym, where 0 = completely incorrect and 1 = fully correct (i.e. higher scores mean a better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Opeolu Adeoye, MD, Study Chair — Washington University School of Medicine
Locations (1):
- American Heart Association, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No